Comprehensive Cancer Center of Wake Forest University (CCCWFU)

**CCCWFU 99516** 

**Principal Investigator:** John M. Salsman, Ph.D.

Director of Clinical Research in Adolescent and

Young Adult Oncology

Wake Forest School of Medicine

**Co-Investigator(s):** Lynne Wagner, Ph.D.

Professor

Department of Social Sciences and Health Policy

Wake Forest School of Medicine

Judith Moskowitz, Ph.D.

Professor

Department of Medical Social Sciences

Northwestern University Feinberg School of Medicine

Biostatistician: Janet A. Tooze

Comprehensive Cancer Center of Wake Forest

University

Study Coordinator: Denisha Little-Greene, MMS

**Study Recruiter:** 

Protocol Editor: Denisha Little-Greene, MMS

Participating Institution(s): Northwestern University Feinberg School of Medicine

Version Date:03.14.2016Amended:12.15.20166.26.2017

6.30.2017 12.29.17

NCT02832154

Confidential

# Comprehensive Cancer Center of Wake Forest University (CCCWFU) CCCWFU 99516

### **Table of Contents**

| <u>1.0</u> | Introduction and Background | 3 |
|---|---|---|
| <u>2.0</u> | Objectives | 4 |
| <u>3.0</u> | Study Population | 4 |
| <u>4.0</u> | <u>Methods</u> | 5 |
| <u>5.0</u> | Outcome Measures | 7 |
| <u>6.0</u> | Analytic Plan | 8 |
| <u>7.0</u> | Data Managment | 9 |
| <u>8.0</u> | Confidentiality and Privacy | 100 |
| 9.0 | Data Safety and Monitoring | 100 |
| 10.0 | Reporting of Unanticipated Problems, Adverse Events or Deviations | 11 |

Comprehensive Cancer Center of Wake Forest University (CCCWFU)

CCCWFU 99516

### 1.0 Background, Rationale and Context

In preparation for a full-scale randomized clinical trial (RCT) of an internet-delivered positive affect (PA) intervention for young adult cancer survivors, the EMPOWER study will collect pilot data on the feasibility and acceptability of a theoretically-driven, empirically-grounded, individual intervention to promote positive affect (PA). An innovative, intervention for HIV patients (Lessons in Linking Affect and Coping: LILAC) will be adapted for use with young adult cancer survivors. This intervention teaches eight cognitive and behavioral skills to enhance PA, which may broaden and enhance an individual's resources for adapting to stressful events. Feasibility and acceptability data will be collected with reports of daily positive and negative affect, general and domain-specific health-related quality of life, psychological well-being, and health behaviors. This will provide data to support further intervention studies, including an R01 proposal of a full-scale randomized clinical trial.

The number of people surviving cancer and even thriving with cancer grows annually. Historically, positive adjustment and growth in cancer has received little attention compared to impairment, disability and psychosocial morbidity. Today, this important area of research is demonstrating increased growth and interest <sup>3,4,5,6,7</sup> with significant potential applications for cancer control and population sciences. <sup>8</sup>

A number of different psychosocial interventions have proven effective with cancer patients. The majority of these interventions are group-based and focus on alleviating the psychosocial burden of cancer by reducing or managing psychological distress. 9-12 Few interventions explicitly target PA. However, such interventions show promise for not only reducing the negative psychosocial impact of cancer and its treatment but for enhancing its positive psychosocial impact as well. 13-16 A potential limiting factor of these PA interventions is that they are primarily group interventions targeted towards advanced cancer patients. Little is known about individualized PA interventions for cancer patients or survivors, but emerging and innovative research of a PA intervention for newly diagnosed HIV patients<sup>17-18</sup> may have applications for cancer patients. Guided by Fredrickson's broaden-and-build theory of positive emotions<sup>22</sup> and funded by the NIMH (R01MH084723), Moskowitz's RCT of a 5-session evidence-based intervention is designed to teach skills for increasing the frequency and intensity of daily PA and to examine the intervention's effects on subsequent psychological well-being. health behaviors, and physical health after diagnosis with HIV. Patients with HIV experience similar negative and positive psychosocial seguelae as patients with cancer. 19-22 This manualized web-based and home-delivered intervention (LILAC) focused explicitly on increasing positive affect, and has shown good feasibility, acceptability, and preliminary efficacy in people coping with significant healthrelated stress <sup>23,24</sup> including women with advanced breast cancer. Thus. Moskowitz' empirically-based PA intervention research may have beneficial

Comprehensive Cancer Center of Wake Forest University (CCCWFU)

CCCWFU 99516

parallels to inform this current project. In this application, we propose to build on this prior work to adapt the LILAC intervention to improve health-related quality of life (HRQOL) for young adult survivors of cancer.

### 2.0 Objectives

- 2.1 Primary Objectives
  - 2.1.1 To adapt an individualized positive affect intervention that was developed for newly diagnosed HIV patients to use with young adult cancer survivors.
  - 2.1.2 To pilot test the positive affect intervention with young adult cancer survivors to determine its feasibility and acceptability.
- 2.2 Secondary Objective
  - 2.2.1 To describe health related quality of life, psychological well-being, and health behaviors in young adult cancer survivors

### 3.0 Study Population

60 young adult cancer survivors will be recruited through the Comprehensive Cancer Center of Wake Forest University (N=40) and the Robert H. Lurie Comprehensive Cancer Center of Northwestern University (N=20).

All patients will meet the following inclusion criteria:

- Able to read and understand English
- Past history of a cancer diagnosis (excluding basal cell skin carcinoma)
- 15 to 39 years of age at diagnosis of first cancer and currently between the ages of 18-39
- Within 0-5 years post-active treatment for initial diagnosis or recurrence
- Wireless internet connection or a home computer that is connected to the internet

#### Exclusion criteria:

- Currently receiving palliative or hospice care
- Significant psychiatric history

We anticipate a large percentage of our target sample to have active mywakehealth accounts, and we plan to use the secure MyChart portal to send study information to potentially eligible patients to gauge their interest in the study and communicate as necessary with consented participants.

Comprehensive Cancer Center of Wake Forest University (CCCWFU)

CCCWFU 99516

#### 4.0 Methods

#### 4.1 Registration Procedures

All patients entered on any CCCWFU trial, whether treatment, companion, or cancer control trial, **must** be registered with the CCCWFU Protocol Registrar or entered into ORIS Screening Log within 24 hours of Informed Consent. Patients **must** be registered prior to the initiation of treatment.

You must perform the following steps in order to ensure prompt registration of your patient:

- 1. Complete the Eligibility Checklist (Appendix B)
- 2. Complete the Protocol Registration Form (Appendix A)
- 3. Alert the Cancer Center registrar by phone, *and then* send the signed Informed Consent Form, Eligibility Checklist and Protocol Registration Form to the registrar, either by fax or e-mail.

\*Protocol Registration is open from 8:30 AM - 4:00 PM, Monday-Friday.

4. Fax/e-mail ALL eligibility source documents with registration. Patients will not be registered without all required supporting documents.

Note: If labs were performed at an outside institution, provide a printout of the results. Ensure that the most recent lab values are sent.

To complete the registration process, the Registrar will:

- assign a patient study number
- register the patient on the study

#### 4.2 Study Design

Patients will be recruited through RHLCCC and CCCWFU. Study staff will work with the Wake Forest Health Sciences Comprehensive Cancer Center's Cancer Informatics Group to identify potential CCCWFU patients from the electronic medical record and/or cancer registry. Potentially eligible patients will be recruited through a direct in-clinic approach as well as mailed letters followed by a phone call by a study team member. The recruitment call will be followed by an email

Comprehensive Cancer Center of Wake Forest University (CCCWFU)

CCCWFU 99516

outlining the details discussed during the phone call and instructions on next steps and a link to the screening questionnaire (*Recruitment Email Script*). IRB-approved study flyers will be placed in the community at large, the Comprehensive Cancer Center at Wake Forest Baptist Medical Center and other strategic locations associated with Wake Forest Baptist Medical Center. IRB-approved study flyers may also be disseminated through email blasts or postings on websites of local cancer support agencies such as Cancer Services.

Patients will then be screened for eligibility using an online screening questionnaire on Qualtrics. Those that are ineligible will be displayed a message stating that he/she was ineligible. Patients who are eligible based will be navigated to the consent form and initial study questionnaire on Qualtrics, an online data collection tool that enables researchers to create study-specific websites for capturing patient data securely online. The instrument library includes self-report batteries or profiles from Patient-Reported Outcomes Measurement Information System (PROMIS) and the NIH Toolbox which include many of the measures that will be used in the study. At completion of the baseline questionnaire, all patients will be given access to the PA intervention.

The PA intervention is a 5 session online intervention that teaches 8 skills for increasing the frequency of positive emotions: 1) noting daily positive events<sup>25-28</sup> 2) capitalizing on or savoring positive events;<sup>29-30</sup> 3) gratitude;<sup>31-33</sup> 4) mindfulness;<sup>34-37</sup> 5) positive reappraisal;<sup>38-45</sup> 6) focusing on personal strengths;<sup>42-43,49-52</sup> 7) setting and working toward attainable goals;<sup>53-54,55-58</sup> and 8) small acts of kindness.<sup>59-63</sup> The skills are presented over the course of 5 weeks. A week will consist of 1-2 days of didactic material and several days of brief, real-life skills practice and reporting, with each day's "home practice" taking approximately 20-30 minutes to complete. Patients cannot skip ahead, but they can return to old lessons or exercises if they choose. Most exercises are done in a "diary" format in which patients' past responses are displayed next to their new ones, so that every time the patient visits that exercise they see their growing list of past positive experiences. Patients will be permitted up to 8 weeks to complete this self-guided intervention to account for normal interruptions and unexpected delays in life.

Acceptability Interview. Research staff will conduct a 30-minute audio-recorded, post-intervention phone interview with all patients approximately one week after the intervention is complete to gather acceptability data. The semi-structured interview includes questions where participants rank the skill sessions in terms of favorite topics, the likelihood of referral to others (a friend or someone diagnosed with cancer) and the likelihood of practicing learned skills. There is also a section with open-ended questions, including questions about participant experiences with use of the website and home practice exercises

Patient Incentives. Each patient will be paid \$10 for each completed assessment for a maximum of \$30. Patients will be paid in full upon completion of the study via virtual gift card.

Comprehensive Cancer Center of Wake Forest University (CCCWFU)

CCCWFU 99516

Fidelity Monitoring. Whether patients understood and remember the intervention content will be assessed via multiple-choice "quiz" questions within each lesson. If patients are not able to answer a question, it will trigger a review of the relevant material (patients can also choose to review past material at any time). How frequently patients visit the website and how many times they complete the daily practice exercises for each skill will also be recorded. This information can be used in "dose-response" analyses to determine whether greater exposure to the exercises leads to stronger intervention effects. Patient progress will be monitored during the study and patients who appear to be having trouble or are disengaging from the intervention will be contacted. Our experience indicates that even very brief human contact can increase patients' commitment to the intervention. Patients will receive an email or phone call from a study staff member if they fail to visit the website more than 3 days in a week. Patients who cannot be reached or who do not resume visiting the website but also don't ask to leave the study will be re-contacted once per week for 3 weeks. After that they will be counted as noncompleters, though we will still try to contact them to obtain post-intervention measures. Patients who do not reach the final lesson at the end of 8 weeks will also be considered non-completers and will be asked to take the post-intervention measures at that time.

#### 5.0 Study Outcomes and Study Measures

Patients will complete self-report questionnaires at baseline (pre-test), approximately 8 weeks after baseline (post-test), then at 12 weeks (follow-up) for a total of 3 assessments, each lasting approximately 25-30 minutes. All measures will be completed from home via patients' personal computers. In addition to the measures listed below, key demographics will be assessed (race/ethnicity, education, household income, insurance status), cancer type, time since diagnosis, type of treatment, and time since treatment (See Appendix 3 for a complete list of measures).

#### 5.1 Primary Outcomes

The primary outcomes for this study are measures of feasibility – accrual, refusal, retention, adherence and acceptability.

#### 5.2 Secondary Outcomes

**5.2.1** Health-Related Quality of Life (HRQOL). The PROMIS global health items will be used to assess overall HRQOL, 68 and the PROMIS-2969-70 to assess domain-specific aspects of HRQOL. The PROMIS Global scale consists of 10 items that assess general health, including overall physical and mental health. The PROMIS-29 consists of 29 items that assess physical functioning, anxiety, depression, fatigue, sleep disturbance, social

Comprehensive Cancer Center of Wake Forest University (CCCWFU)

CCCWFU 99516

functioning, pain interference, and pain intensity. These PROMIS measures will be supplemented with additional items from the PROMIS physical function short form<sup>71</sup> and the PROMIS anger short form.<sup>72</sup> The 4 PROMIS items for depression in this measure do not assess suicidality.

- **5.2.2** Psychological well-being. Psychological well-being will be assessed with NIH Toolbox short forms for positive affect, life satisfaction, and meaning and purpose. In addition, the NIH PROMIS General Self-Efficacy short form will be administered as it is a closely related construct to psychological well-being and positively associated with better patient-reported outcomes.
- **5.2.3** *Health Behaviors.* Healthy behaviors often associated with enhanced coping and better adjustment will be assessed. Physical health behaviors will include: diet, exercise, alcohol consumption, and cigarette smoking.

#### 6.0 Statistical Considerations

Wake Forest School of Medicine will be the Coordinating Center for the study and will conduct all data analysis.

#### 6.1 Analysis of Primary Objective

Accrual will be estimated as the number of patients accrued divided by the number of months of accrual. A 95% confidence interval for the monthly accrual rate will be calculated based on the Poisson distribution. The refusal rate will be estimated as the number of patients who refuse to participate divided by the number eligible. Retention will be primarily defined as the proportion of patients who provide 8 week and 12 week data. Patients who discontinue the intervention (refuse phone calls) but complete the outcome assessments will be counted in the numerator for calculating retention. Retention estimates will be calculated overall and by site. Adherence to the intervention will be calculated as the number of intervention sessions completed, the frequency of completing exercises, and number of website visits. We will calculate and report the mean adherence across all individuals as well as the proportion of patients who completed three or more sessions. Several measures will be used to quantify acceptability, including quantitative measures and interview. Means and the proportion responding affirmatively to the highest two responses for each question will be combined and exact 95% CIs will be calculated for these estimates. In addition, Dr. Salsman and Dr. Moskowitz will review open-ended (written) feedback and audio-recordings of phone interviews to identify meta-themes and determine saturation of concepts.<sup>78</sup>

Comprehensive Cancer Center of Wake Forest University (CCCWFU)

CCCWFU 99516

#### 6.2 Analysis of Secondary Objective

Quantitative outcomes will be assessed by a covariance pattern model for repeated measures to examine change in PA and PROMIS scores over time.

#### 6.2 Power and Sample Size

While this is a pilot study and we will not be testing the efficacy of the intervention, we do want to be able to estimate feasibility, acceptability, and changes in PA and PROMIS scores with a fair degree of precision. With a total of 60 patients we can estimate confidence intervals around means to within ±0.25 SD, and proportions within ±12.7%, with 95% confidence. Assuming that 20% of the patients may drop out, we could estimate confidence intervals for means within ±0.28 SD and proportions within ±14.1% for measures evaluated at the end of the study. Furthermore, the sample size of N=60 should permit us to achieve data saturation, or the point at which successive information serves only to replicate previous content themes and no new information is obtained.<sup>79</sup> Past research reveals that saturation often occurs within the first 12 interviews.<sup>78</sup>

#### 6.3 Estimated Accrual Rate

It is anticipated that 3.2 patients a month will be accrued to this trial, meeting the target of 60 in 19 months. To date, we have recruited 18 patients in 6 months at the Robert H. Lurie Comprehensive Cancer Center of Northwestern University.

#### 6.4 Estimated Study Length

Patients will complete their participation in 12 weeks, for an estimated study length of 15 months.

### 7.0 Data Management

The web intervention is delivered via a customized website built on Moodle, a courseware platform that is used by schools and universities worldwide. Moodle allows delivery of text or video instruction as well as interactive activities such as journals and adaptive quizzes. Moodle is recognized as secure and well-tested software, and HIPAA-compliant. All communications with the website will use industry-standard TLS/SSL encryption. Another layer of security will be provided by avoiding any use of personally identifiable information, medical information, or other sensitive information in the context of the intervention. Patients' Moodle accounts will not be linked to their real name or email address. The design of our intervention website has been refined through a number of iterations based on user testing and feedback from study patients (e.g., simplifying the interface,

Comprehensive Cancer Center of Wake Forest University (CCCWFU)

CCCWFU 99516

clearly labeling new material and exercises). We have also ensured that material is viewable on handheld, tablet, and laptop devices.

| Informed consent document | ORIS |
|---|---|
| Protocol registration form | ORIS |
| Pre-, post- and follow-up test | Qualtrics |
| Questionnaires (Qualtrics) | |
| Intervention Sessions 1-5 | Moodle |
| Phone Interview | Audio-recorded and stored among password protected study files |

### 8.0 Confidentiality and Privacy

Confidentiality will be protected by collecting only information needed to assess study outcomes, minimizing to the fullest extent possible the collection of any information that could directly identify subjects, and maintaining all study information in a secure manner. To help ensure subject privacy and confidentiality, only a unique study identifier will appear on the data collection form. Any collected patient identifying information corresponding to the unique study identifier will be maintained on a linkage file, store separately from the data. The linkage file will be kept secure, with access limited to designated study personnel. Following data collection subject identifying information will be destroyed (state the anticipated time the data will be destroyed, e.g. three years after closure of the study, and the method of destruction), consistent with data validation and study design, producing an anonymous analytical data set. Data access will be limited to study staff. Data and records will be kept locked and secured, with any computer data password protected. No reference to any individual patient will appear in reports, presentations, or publications that may arise from the study.

### 9.0 Data Safety and Monitoring

The principal investigator will be responsible for the overall monitoring of the data and safety of study patients. The principal investigator will be assisted by other members of the study staff.

The risks of this study are low; however staff will be trained to handle situations with sensitivity and empathy. The study coordinator will be trained to monitor for significant patient distress or depressive symptoms and will be instructed on the appropriate courses of referral is a patient is considered to be at risk for a safety concern.

Comprehensive Cancer Center of Wake Forest University (CCCWFU)

CCCWFU 99516

# **10.0** Reporting of Unanticipated Problems, Adverse Events or Deviations

Any unanticipated problems, serious and unexpected adverse events, deviations or protocol changes will be promptly reported by the principal investigator or designated member of the research team to the IRB and sponsor or appropriate government agency if appropriate.

## Comprehensive Cancer Center of Wake Forest University (CCCWFU) CCCWFU 99516

#### References

- 1. Moskowitz JT. Coping interventions and the regulation of positive affect. In: Folkman S, ed. The Oxford handbook of stress, health, and coping. Oxford; New York: Oxford University Press; 2011.
- 2. Fredrickson BL. The role of positive emotions in positive psychology. The broaden-and-build theory of positive emotions. Am. Psychol. 03 2001;56(3):218-226.
- 3. Aspinwall LG, Tedeschi RG. The Value of Positive Psychology for Health Psychology: Progress and Pitfalls in Examining the Relation of Positive Phenomena to Health. *Ann. Behav. Med.* 2010;39(1):4-15.
- **4.** Aspinwall LG, Tedeschi RG. Of Babies and Bathwater: A Reply to Coyne and Tennen's Views on Positive Psychology and Health. *Ann. Behav. Med.* 2010;39(1):27-34.
- **5.** Coyne JC, Ranchor AV. Positive Psychology in Cancer Care: A Story Line Resistant to Evidence. *Ann. Behav. Med.* 2010;39(1):35-42.
- 6. Coyne JC, Tennen H. Positive Psychology in Cancer Care: Bad Science, Exaggerated Claims, and Unproven Medicine. *Ann. Behav. Med.* 2010;39(1):16-26.
- 7. Miller SM, Sherman AC, Christensen AJ. Introduction to Special Series: The Great Debate--Evaluating the Health Implications of Positive Psychology. *Ann. Behav. Med.* 2010;39(1):1-3.
- **8.** Gorin SS. Theory, Measurement, and Controversy in Positive Psychology, Health Psychology, and Cancer: Basics and Next Steps. *Ann. Behav. Med.* 2010;39(1):43-47.
- 9. Meyer TJ, Mark MM. Effects of psychosocial interventions with adult cancer patients: a meta-analysis of randomized experiments. Health Psychol. 1995;14(2):101-108.
- 10. Newell SA, Sanson-Fisher RW, Savolainen NJ. Systematic Review of Psychological Therapies for Cancer Patients: Overview and Recommendations for Future Research. J. Natl. Cancer Inst. 2002;94(8):558-584.
- 11. Rehse B, Pukrop R. Effects of psychosocial interventions on quality of life in adult cancer patients: meta analysis of 37 published controlled outcome studies. Patient Educ. Couns. 2003;50(2):179-186.
- 12. Sheard T, Maguire P. The effect of psychological interventions on anxiety and depression in cancer patients: results of two meta-analyses. Br. J. Cancer. 1999;80(11):1770-1780.
- 13. Breitbart W. Spirituality and meaning in supportive care: spirituality and meaning-centered group psychotherapy interventions in advanced cancer. Support. Care Cancer. 2002;10(4):272-280.
- 14. Ramachandra P, Booth S, Pieters T, Vrotsou K, Huppert FA. A brief self-administered psychological intervention to improve well-being in patients with cancer: Results from a feasibility study. Psychooncology. 2009;18(12):1323-1326.
- 15. Lee V, Cohen SR, Edgar L, Laizner AM, Gagnon AJ. Meaning-making and psychological adjustment to cancer: development of an intervention and pilot results. Oncol. Nurs. Forum. Mar 2006;33(2):291-302.
- 16. Chochinov HM, Hack T, Hassard T, Kristjanson LJ, McClement S, Harlos M. Dignity Therapy: A Novel Psychotherapeutic Intervention for Patients Near the End of Life. J. Clin. Oncol. 2005;23(24):5520-5525.
- 17. Moskowitz JT. Coping interventions and the regulation of positive affect. In: Folkman S, ed. The Oxford handbook of stress, health, and coping. Oxford; New York: Oxford University Press; 2011.
- 18. Moskowitz JT. Positive affect at the onset of chronic illness: planting the seeds of resilience. In: Reich JW, Zautra A, Hall JS, eds. Handbook of adult resilience. New York: Guilford Press; 2010.
- 19. Fredrickson BL. The role of positive emotions in positive psychology. The broaden-and-build theory of positive emotions. Am. Psychol. 03 2001;56(3):218-226.
- 20. Sherman AC, Mosier J, Leszcz M, et al. Group Interventions for Patients with Cancer and HIV Disease: Part I: Effects on Psychosocial and Functional Outcomes at Different Phases of Illness. Int. J. Group Psychother. 2004;54(1):29.

## Comprehensive Cancer Center of Wake Forest University (CCCWFU) CCCWFU 99516

- 21. Lechner S, Weaver K. Lessons learned about benefit finding among individuals with cancer of HIV/AIDS. In: Park CL, American Psychological Association, eds. Medical illness and positive life change: can crisis lead to personal transformation? Washington, DC: American Psychological Association; 2009:185-206.
- 22. Sawyer A, Ayers S, Field AP. Posttraumatic growth and adjustment among individuals with cancer or HIV/AIDS: A meta-analysis. Clin. Psychol. Rev. 2010;30(4):436-447.
- 23. Moskowitz JT, Hult JR, Duncan LG, et al. A Positive Affect Intervention for People Experiencing Health-Related Stress: Development and Non-Randomized Pilot Test. *J Health Psychol*. October 21, 2011 2012;17(5):677-693.
- 24. Saslow LR, Cohn M, Moskowitz JT. Positive Affect Interventions to Reduce Stress: Harnessing the Benefit while Avoiding the Pollyanna. In: Gruber J, Moskowitz JT, eds. *The Dark and Light Sides of Positive Emotion*. New York: Oxford University Press; 2014:515-532.
- **25.** Krause N. Positive life events and depressive symptoms in older adults. Behavioral Medicine. 1998;14(101-112).
- **26.** Lewinsohn PM, Hoberman HM, Clarke GN. The coping with depression course: Review and future directions. Canadian Journal of Behavioral Science. 1989;21:470-493.
- 27. Lewinsohn PM, Amenson CS. Some relations between pleasant and unpleasant mood-related events and depression. Journal of Abnormal Psychology. 1978;87:644-654.
- **28.** Lewinsohn PM, Sullivan M, Grosscup SJ. Changing reinforcing events: An approach to the treatment of depression. Psychotherapy: Theory, research, and practice. 1980;17:322-334.
- **29.** Langston CA. Capitalizing on and coping with daily-life events: Expressive responses to positive events. Journal of Personality and Social Psychology. 1994;67:1112-1125.
- **30.** Bryant FB. A four-factor model of perceived control: Avoiding, coping, obtaining, and savoring. Journal of Personality. 1989;57:773-797.
- **31.** Emmons RA. Thanks! how the new science of gratitude can make you happier. New York: Houghton Mifflin; 2007.
- **32.** Kashdan TB, Uswatte G, Julian T. Gratitude and hedonic and eudaimonic well-being in Vietnam war veterans. Behaviour Research and Therapy. 2006;44:177-199.
- **33.** Lyubomirsky S, Sheldon K, Schkade D. Pursuing happiness: The architecture of sustainable change. Review of General Psychology. 2005;9:111-131.
- 34. Kabat-Zinn J. Mindfulness-Based interventions in context: Past, present, and future. Clinical Psychology: Science and Practice. 2003;10:144-156.
- 35. Grossman P, Tiefenthaler-Gilmer U, Raysz A, Kesper U. Mindfulness training as an intervention for fibromyalgia: Evidence of postintervention and 3-year follow-up benefits in well-being. Psychotherapy and Psychosomatics. 2007;76:226-233.
- 36. Shapiro M, Brown KW, Biegel GM. Teaching self-care to caregivers: Effects of mindfulness-based stress reduction on the mental health of therapists in training. Training and Education in Professional Psychology. 2007;1:105-115.
- 37. Cresswell JD, Myers HF, Cole SW, Irwin MR. Mindfulness meditation training effects on CD4+ T lymphocytes in HIV-1 infected adults: A small randomized controlled trial. Brain Behavior and Immunity. 2009;23:184-188.
- **38.** Folkman S. Positive psychological states and coping with severe stress. Social Science and Medicine.1997;45:1207-1221.
- 39. Sears SR, Stanton AL, Danoff-Burg S. The yellow brick road and the emerald city: Benefit finding, positive reappraisal coping and posttraumatic growth in women with early-stage breast cancer. Health Psychology. Sep 2003:22(5):487-497.
- **40.** Carver CS, Scheier MF. Situational coping and coping dispositions in a stressful transaction. Journal of Personality and Social Psychology. 1994;66:184-195.
- 41. Moskowitz JT, Folkman S, Collette L, Vittinghoff E. Coping and mood during AIDS-related

## Comprehensive Cancer Center of Wake Forest University (CCCWFU) CCCWFU 99516

- caregiving and bereavement. Annals of Behavioral Medicine. 1996;18(1):49-57.
- 42. Moskowitz JT, Hult JR, Bussolari C, Acree M. What works in coping with HIV? A meta-analysis with implications for coping with serious illness. Psychological Bulletin. Jan 2009;135(1):121-141.
- 43. Antoni MH, Ironson G, Schneiderman N. Cognitive-behavioral stress management for individuals living with HIV. New York: Oxford University Press; 2007.
- 44. Chesney M, Chambers D, Taylor JM, Johnson LM, Folkman S. Coping effectiveness training for men living with HIV: Results from a randomized clinical trial testing a group-based intervention. Pyschosomatic Medicine. 2003;65:1038-1046.
- 45. Chesney MA, Folkman S, Chambers D. Coping effectiveness training. International Journal of STD and AIDS. 1996;7 (Suppl. 2):75-82.
- **46.** Koole SL, Smeets K, van Knippenberg A, Dijksterhuis A. The cessation of rumination through self- affirmation. Journal of Personality and Social Psychology. 1999;77:111-125.
- 47. Taylor SE, Kemeny ME, Aspinwall LG, Schneider SG, Rodriguez R, Herbert M. Optimism, coping, psychological distress, and high-risk sexual behavior among men at risk for Acquired Immunodeficiency Syndrome (AIDS). Journal of Personality and Social Psychology. 1992;63:460-473.
- **48.** Taylor SE, Lobel M. Social comparison activity under threat: Downward evaluation and upward contacts. Psychological Review. 1989;96:569-575.
- **49.** Carver CS, Scheier MF. Origins and functions of positive and negative affect: A control process view. Psychological Review. 1990;97:19-35.
- 50. Lent RW, Singley D, Sheu H-B, et al. Social cognitive predictors of domain and life satisfaction: Exploring the theoretical precursors of subjective well-being. J Consult Clin Psychol. 2005:52:429-442.
- 51. Sikkema KJ, Kalichman SC, Kelly, J.A., Koob JJ. Group intervention to improve coping with AIDS- related bereavement: Model development and an illustrative clinical example. AIDS Care. 1995;7:463-475.
- 52. Brunstein JC, Schultheiss OC, Grassmann R. Personal goals and emotional well-being: The moderating role of motive dispositions. Journal of Personality and Social Psychology. 1998;75(2):494-508.
- Moskowitz JT, Hult JR, Bussolari C, Acree M. What works in coping with HIV? A meta-analysis with implications for coping with serious illness. Psychological Bulletin. Jan 2009;135(1):121-141.
- **54.** Antoni MH, Ironson G, Schneiderman N. Cognitive-behavioral stress management for individuals living with HIV. New York: Oxford University Press; 2007.
- 55. Carver CS, Scheier MF. Origins and functions of positive and negative affect: A control process view. Psychological Review. 1990;97:19-35.
- **56.** Lent RW, Singley D, Sheu H-B, et al. Social cognitive predictors of domain and life satisfaction: Exploring the theoretical precursors of subjective well-being. J Consult Clin Psychol. 2005;52:429-442.
- 57. Sikkema KJ, Kalichman SC, Kelly, J.A., Koob JJ. Group intervention to improve coping with AIDS- related bereavement: Model development and an illustrative clinical example. AIDS Care. 1995;7:463-475.
- 58. Brunstein JC, Schultheiss OC, Grassmann R. Personal goals and emotional well-being: The moderating role of motive dispositions. Journal of Personality and Social Psychology. 1998;75(2):494-508.59. Musick MA, Wilson J. Volunteering and depression: the role of psychological and social resources in different age groups. Soc Sci Med. 2003;56:259-269.
- 60. Oman D, Thoresen CE, McMahon K. Volunteerism and mortality among the community-dwelling elderly. J Health Psychol. 1999;4:301-316.
- 61. Moen P, Dempster-McCain D, Williams RM. Successful aging. American Journal of Sociology.

## Comprehensive Cancer Center of Wake Forest University (CCCWFU) CCCWFU 99516

1993;97:1612- 1632.

- **62.** Penner LA, Dovidio JF, Piliavin JA, Schroeder DA. Prosocial behavior: Multilevel perspectives. Annu Rev Psychol. 2005;56:365-392.
- 63. Brown SL, Nesse RM, Vinokur AD, Smith DM. Providing social support may be more beneficial than receiving it: Results from a prospective study of mortality. Psychol Sci. 2003;14:320-327.
- 64. Cole-Lewis H, Kershaw T. Text messaging as a tool for behavior change in disease prevention and management. Epidemiologic reviews. 2010;32(1):56-69.
- **65.** Fogg BJ, Adler R. Persuasive Technology L. Texting 4 health: a simple, powerful way to improve lives. Stanford, CA: Stanford University; 2009.
- 66. Fry JP, Neff RA. Periodic prompts and reminders in health promotion and health behavior interventions: systematic review. Journal of medical Internet research. 2009;11(2).
- Baumeister RF, Vohs KD. Self-Regulation, ego depletion, and motivation. Social and Personality Psychology Compass. 2007;1(1):115-128.
- 68. Hays RD, Bjorner JB, Revicki DA, Spritzer KL, Cella D. Development of physical and mental health summary scores from the patient-reported outcomes measurement information system (PROMIS) global items. Quality of Life Research. 2009;18(7):873-880.
- 69. Beaumont JL, Cella D, Phan AT, et al: Comparison of Health-Related Quality of Life in Patients With Neuroendocrine Tumors With Quality of Life in the General US Population. Pancreas 41:461-466, 2012.
- 70. Hinchcliff M, Beaumont JL, Thavarajah K, et al: Validity of two new patient-reported outcome measures in systemic sclerosis: Patient-reported outcomes measurement information system 29-item health profile and functional assessment of chronic illness therapy—dyspnea short form. Arthritis Care and Research 63:1620-1628, 2011
- 71. Fries, J. F., Cella, D., Rose, M., Krishnan, E., Bruce, B. (2009). Progress in assessing physical function in arthritis: PROMIS short forms and computerized adaptive testing. Journal of Rheumatology, 36(9), 2061-6. (PMCID: Pending)
- 72. Pilkonis, P. A., Choi, S. W., Reise, S. P., Stover, A. M., Riley, W. T., & Cella, D. (2011). Item banks for measuring emotional distress from the Patient-Reported Outcomes Measurement Information System (PROMIS<sup>TM</sup>): Depression, anxiety, and anger. Assessment, 18(3), 263-283. (PMCID: PMC3153635)
- 73. Salsman, J.M., Lai, J-S, Hendrie, H.C., Butt, Z., Zill, N., Pilkonis, P.A., Peterson, C., Stoney, C.M., Brouwers, P., & Cella, D. Assessing psychological well-being: Self-report instruments for the NIH Toolbox. Quality of Life Research. 2013; 23(1):205-15
- 74. Kupst MJ, Butt Z, Stoney CM, Griffith JW, Salsman JM, Folkman S, Cella D. Assessment of Stress and Self- Efficacy for the NIH Toolbox for Neurological and Behavioral Function. Anxiety, Stress, & Coping. 2015; Jan. 12 [Epub ahead of print]
- 75. Doyle C, Kushi LH, Byers T, et al.: Nutrition and physical activity during and after cancer treatment: An American Cancer Society Guide for Informed Choices. CA Cancer J Clin, Nov 2006; 56: 323 353.
- 76. Hesse, Bradford, and Richard Moser. Health Information National Trends Survey (HINTS), 2007. ICPSR25262- v1. Ann Arbor, MI: Inter-university Consortium for Political and Social Research [distributor], 2009-06-23. http://doi.org/10.3886/ICPSR25262.v1
- 77. Godin G Shephard RJ. A simple method to assess exercise behavior in the community. Can J Applied Sport Sciences. 1985; 10: 141-146.
- **78.** Guest G, Bunce A, Johnson L. How Many Interviews Are Enough? An Experiment with Data Saturation and Variability. *Field Meth.* 2006;18(1):59-82.
- **79.** Bowen GA. Naturalistic inquiry and the saturation concept: a research note. *Qualitative research: QR* 2008;8(1):137-152.

Comprehensive Cancer Center of Wake Forest University (CCCWFU) CCCWFU 99516

### Appendix A – Subject Eligibility Checklist

| IRB Protocol No. | CCCWFU Proto | ocol No. | | | |
|---|---|---|---|---|---|
| Study Title: | | | | | |
| Principal Investigator: | | | | | |
| Inclusion Criteria<br>(as outlined in study pro | | Criteria<br>is met | Criteria is NOT met | (Plea | Source Used to Confirm * use document dates and lab results) |
| Exclusion Criteria<br>(as outlined in study pro | | Criteria<br>NOT<br>present | Criteria is present | (Plea | Source Used to Confirm * use document dates and lab results) |
| This subject is eligible / | ineligible for | r participa | tion in this st | tudy. | |
| ORIS Assigned PID: | | | | | |
| Signature of research profession | al confirming el | igibility: | | | Date: |
| Signature of Treating Physician* | *.<br> | | | | Date: |

<sup>\*</sup> Examples of source documents include clinic note, pathology report, laboratory results, etc. When listing the source, specifically state which document in the medical record was used to assess eligibility. Also include the date on the document. Example: "Pathology report, 01/01/14" or "Clinic note, 01/01/14"

<sup>\*\*</sup>Principal Investigator signature can be obtained following registration if needed

Comprehensive Cancer Center of Wake Forest University (CCCWFU)

CCCWFU 99516

#### APPENDIX B: REDUCED REGISTRATION FORM

# Comprehensive Cancer Center of Wake Forest University REDUCED REVIEW\*\* REGISTRATION FORM

| Protocol #: | | _ | | | *Required Fields |
|---|---|---|---|---|---|
| Protocol Title:<br>(optional) | | | | | |
| DEMOGRAPHICS | | | | | |
| Name (last, first):<br>(or initials) | | | | _ | |
| (or initials), | | (required if no MRN | | | |
| *SEX O MALE | ○ FEMA | ALE. | | | |
| *ETHNICITY (choose one): | O HISPA | ANIC | O NON-HIS | SPANIC | |
| *RACE (choose all that apply): | □ WHIT | TE [ | AFRICA | N-AMERICAN | |
| | ASIA | N [ | PACIFIC | C ISLANDER (HAWAIIAN) | ) |
| | NATI | IVE AMERICA | N (ALASKA | AN) | |
| *DIAGNOSIS: | | | | | |
| BIRTH DATE: | (i | include if no N | IRN is provi | ded) | |
| *MD Name (last, first): | | | | | |
| *DATE CONSENT WAS SIGNE | ED | | | | |
| Date of Registration (if differ | ent) | | | | |
| PID #: | (to be cor | mpleted by Re | egistrar) | | |
| The Comprehensive Cancer Ce<br>Registrar the day the patient is<br>communicated to the Centralize | consented; | ; if this is not p | ossible we | require that all registration | |
| **Reduced review means eligib | ility and oth | her review are | not perforn | ned by CRM registrar. | |
| Questions: call 713-6767 | | | | | |
| | Submit | t by Email*** | Prin | nt Form | |

<sup>\*\*\*</sup>If not using the full wfubmc.edu outlook client (full outlook, not web outlook), save this file and attach to an email to registra@wfubmc.edu

Submitter of this form is responsible for insuring that all regulatory and eligibility requirements are met for this registration.

### **Appendix C – Study Measures**

| Variables | Construct/Measures |
|---|---|
| Demographics | Age, gender, ethnic, edu, income, job & mar. status, insurance, etc. |
| Clinical | Cancer dx, stage, adj. tx, etc. |
| Quality of Life | Global Impact Items PROMIS PROMIS Global 10 PROMIS-29 + 4 additional PROMIS physical function items PROMIS Anger SF |
| Psychological<br>Well-Being | NIH PROMIS General Sell-Efficacy Scale SF NIH Toolbox Life Satisfaction SF NIH PROMIS Meaning & Purpose SF NIH Toolbox Positive Affect SF |
| Health<br>Behaviors | Diet Alcohol Use & Smoking Leisure Time Exercise Questionnaire |

### **EMPOWER Sociodemographic Questions**

| SDC01 | What is your current age? | | |
|---|---|---|---|
| SDC02 | Are you of Hispanic origin, such as Lati | n American, | , Mexican, Puerto Rican, or Cuban? |
| | | 01 | Yes, of Hispanic origin |
| | | 02 | No, not of Hispanic origin |
| | | 09 | Decline to answer |
| SDC03 | Do you consider yourself? | | |
| | | 01 | White or Caucasian |
| | | 02 | Black or African American |
| | | 03 | Asian |
| | | 04 | Native Hawaiian/Other Pacific Islander |
| | | 05 | Native American or Alaska Native |
| | | 06 | Mixed racial background |
| | | 07 | Other race |
| | | 09 | Decline to answer |
| SDC04 | What is your gender? | 01 | Female |
| | | 02 | Male |
| SDC05 | What is your marital status? | | |
| | , | 01 | Single, never married |
| | | 02 | Married |
| | | 03 | Divorced |
| | | 04 | Separated |
| | | 05 | Widowed |
| | | 06 | Living with partner |
| SDC06 | Do you currently live alone or with ot | hers? | |
| | , | 01 | Live alone |
| | | 02 | Live with others (e.g., parent, roommate, |
| | | | spouse/partner, brother, sister, children) |
| SDC07 | Are you now responsible for raising an | • | <del>-</del> |
| | | 01 | No |
| | | 02 | Yes |

| SDC08 taxes? | Which of the following income categories | best describes your total household income before |
|---|---|---|
| | 01 | Less than \$15,000 |
| | 02 | \$15,000 to \$24,999 |
| | 03 | \$25,000 to \$34,999 |
| | 04 | \$35,000 to \$49,999 |
| | 05 | \$50,000 to \$74,999 |
| | 06 | \$75,000 to \$99,999 |
| | 07 | \$100,000 to \$124,999 |
| | 08 | \$125,000 to \$149,999 |
| | 09 | \$150,000 to \$199,999 |
| | 10 | \$200,000 to \$249,999 |
| | 11 | \$250,000 or more |
| | 994 | Decline to answer |
| SDC09 | What is the highest level of education you have | e completed? |
| | 01 | Grade school – between 1 and 8 years |
| | 02 | Some high school |
| | 03 | High school diploma or equivalent (e.g., GED) – 12 years |
| | 04 | Some college, vocational or training school |
| | 05 | College graduate |
| | 06 | Some graduate school |
| | 07 | Graduate degree |
| SDC10 | What was your school/employment status <u>right</u> mark all that apply. | t before you were diagnosed with cancer? Please |
| | 01 | Part-time student |
| | 02 | Full-time student |
| | 03 | Working part-time |
| | 04 | Working full-time |
| | 05 | Unemployed |
| | 06 | Full-time homemaker or family caregiver |
| | 07 | Other (please describe in box below) |

| SDC11 | How did your school/employment stamark all that apply. | atus <u>cha</u> i | nge because of your cancer or its treatment? <i>Please</i> |
|---|---|---|---|
| | | 01 | It has not changed because of my cancer or its treatment |
| | | 02 | I quit working completely |
| | | 03 | I quit going to school completely |
| | | 04 | I changed my work status from full-time to part- |
| | | VŦ | time |
| | | 05 | I changed my school status from full-time to part-<br>time |
| | | 06 | I took more than 2 weeks total time off from work |
| | | 07 | I took more than 2 weeks total time off from school |
| | | 08 | Other (please describe in box below) |
| SDC12a | Are you now covered by any type of | of health | insurance? |
| | | 01 | No |
| | | 02 | Yes |
| | Yes, GO TO QUESTION SDC12b<br>SDC12b. How is this health insurar | nce prov | ided? MARK ALL THAT APPLY. |
| | | 01 Th | nrough your employer/school |
| | | 02 Th | nrough your spouse's employer/school |
| | | 03 Th | rough your parent |
| | | | edicaid or other public assistance program |
| | | | ther State Program (for example, Medi-Cal, SCHIP) |
| | | | ilitary or Veteran's Benefits |
| | | 07 Ot | ther (please describe in the box below) |
| | | 09 I d | lon't know |

### **Disease and Treatment Information**

| SDC13 | Please circle which statement best describes your current activity level: | |
|---|---|---|
| | | 0= Normal activity, without symptoms 1= Some symptoms, but do not require bed rest during waking day 2= Require bed rest for less than 50% of waking day 3= Require bed rest for more than 50% of waking day 4= Unable to get out of bed |
| SDC14 | What is your height? (feet/inches) | |
| SDC15 | What is your weight? (lbs) | <u> </u> |
| SDC16 | What was the date of your cancer diagno | osis? (month and year)/ |
| SDC17 | Please select one of the boxes below the your cancer). If none of the boxes is con Basal cell skin cancer Bladder cancer | nt reflects your "primary" cancer diagnosis (e.g., original location of rrect, please select "Other" and explain. Leukemia |
| | Bone tumor | Lung cancer |
| | Brain cancer | ☐ Melanoma (skin cancer) |
| | Breast cancer | ☐ Myeloma |
| | Central Nervous System tumor | ☐ Non-hodgkin lymphoma |
| | Cervical cancer | Ovarian cancer |
| | Colorectal cancer | Prostate cancer |
| | Esophageal cancer | Sarcoma (bone or soft tissue) |
| | Head and neck cancer | ☐ Stomach cancer |
| _<br>bi | Hepatobiliary cancer (liver, pancreas, le duct) | ☐ Testicular cancer |
| | Hodgkin lymphoma | ☐ Thyroid cancer |
| | ] Kidney cancer | Other:(explain) |

| SDC18 Has your cancer spread to any lymph nodes: | |
|---|---|
| | 0=No |
| | 1=Yes |
| | 2=Not sure |
| SDC19a. Has your cancer spread to another part of your bod | y (other than to any lymph nodes)? |
| | 0=No |
| | 1=Yes |
| | 2=Not sure |
| SDC19b. If yes, please check all that apply: | |
| 22 0 15 00 11 you, produce one on the three uppry. | □ Bone |
| | □ Brain |
| | ☐ Lung |
| | □ Liver |
| | ☐ Other: (please specify) |
| SDC20a Are you currently receiving treatment? (check al | l that apply) |
| chemotherapy | |
| radiation treatment | |
| I am not currently receiving treatment. | |
| CDC201 IC 1: 11 1 1:1 | 4 4 16 19 |
| SDC20b If applicable, when did you complete your cance | r treatment(s)? ☐ I did not receive surgery for my cancer. |
| <u> </u> | ☐ I did not receive surgery for my cancer. |
| | ☐ I did not receive enchrotherapy for my cancer |
| c. radiation(month and year) OK | - I did not receive radiation for my cancer |
| SDC21a Where did you receive most of your primary activity radiation therapy)? | e cancer treatment (surgery, chemotherapy, |
| 107 | 01 Academic medical center |
| | 22 Community-based hospital or health center |
| | Office-based private practice |
| SDC21b List the name of the institution where you receive | rad most of your primary active concer |
| treatment (surgery, chemotherapy, radiation therapy). | ed most of your primary active cancer |
| (Surgery, enemotilerapy, radiation therapy). | |
| SDC22 A survivorship care plan (SCP) is a document that it | |
| | g healthy. Following completion of your primary active |
| treatment for cancer, did you receive a SCP from you | |
| | 01 No |
| | 22 Yes |
| | 3 I don't know |
| SDC23 Do you now (within the past month), or have yo | ou ever had any of the following conditions? |
| (please check all that apply) | 2. 2. 2. had any of the following conditions. |

| AIDS/HIV | Hypertension |
|-------------------------|-------------------------|
| Acid Reflux (heartburn) | Insomnia |
| Anemia | Multiple Sclerosis (MS) |
| Anxiety | Migraine/Headaches |
| Arthritis | Ulcers |
| Asthma | Other (specify below) |
| Back Pain | |
| Depression | |
| Diabetes | |
| Fibromyalgia | |
| Heart Disease | |
| Hepatitis | |

### **Global Impact**

| | | Completely<br>positive | Mostly<br>positive; a<br>little negative | A little more positive than negative | Equally<br>positive and<br>negative | A little more<br>negative than<br>positive | Mostly<br>negative;<br>a little<br>positive | Completely<br>negative |
|---|---|---|---|---|---|---|---|---|
| 1 | How positive or negative has the overall impact of your illness been on your views about yourself and your life? | | | 0 | | 0 | | |

| | | Not at all | A little bit | Somewhat | Quite a bit | Very much |
|---|---|---|---|---|---|---|
| 2 | Overall, how much has having your illness affected your views about yourself and your life? | 0 | | 0 | 0 | |

#### Positive Affect

| Positive | Affect | | Positive Affect | |
|---|---|---|---|---|
| | Item ID For the next set of questions, please tell us | | | |
| | | | how true each statement was of you in the past 7 days. | |
| 1 | PA001 | In the past 7 days: | I felt cheerful. | 1 = Not at all 2 = A little bit 3 = Somewhat 4 = Quite a bit 5 = Very much |
| 2 | PA002 | In the past 7 days: | I felt attentive. | 1 = Not at all 2 = A little bit 3 = Somewhat 4 = Quite a bit 5 = Very much |
| 3 | PA006 | In the past 7 days: | I felt delighted. | 1 = Not at all 2 = A little bit 3 = Somewhat 4 = Quite a bit 5 = Very much |
| 4 | PA010 | In the past 7 days: | I felt happy. | 1 = Not at all 2 = A little bit 3 = Somewhat 4 = Quite a bit 5 = Very much |
| 5 | PA014 | In the past 7 days: | I felt joyful. | 1 = Not at all 2 = A little bit 3 = Somewhat 4 = Quite a bit 5 = Very much |
| 6 | PA019 | In the past 7 days: | I felt enthusiastic. | 1 = Not at all 2 = A little bit 3 = Somewhat 4 = Quite a bit 5 = Very much |
| 7 | PA020 | In the past 7 days: | I felt determined. | 1 = Not at all 2 = A little bit 3 = Somewhat 4 = Quite a bit 5 = Very much |
| 8 | PA021 | In the past 7 days: | I felt interested. | 1 = Not at all 2 = A little bit 3 = Somewhat 4 = Quite a bit 5 = Very much |
| 9 | PA025 | In the past 7 days: | I was thinking creatively. | 1 = Not at all 2 = A little bit 3 = Somewhat 4 = Quite a bit 5 = Very much |

| 10 | PA026 | In the past 7 days: | I liked myself. | 1 = Not at all 2 = A little bit 3 = Somewhat 4 = Quite a bit 5 = Very much |
|---|---|---|---|---|
| 11 | PA030 | In the past 7 days: | I felt peaceful. | 1 = Not at all 2 = A little bit 3 = Somewhat 4 = Quite a bit 5 = Very much |
| 12 | PA037 | In the past 7 days: | I felt good-natured. | 1 = Not at all 2 = A little bit 3 = Somewhat 4 = Quite a bit 5 = Very much |
| 13 | PA039 | In the past 7 days: | I felt useful. | 1 = Not at all 2 = A little bit 3 = Somewhat 4 = Quite a bit 5 = Very much |
| 14 | PA042 | In the past 7 days: | I felt understood. | 1 = Not at all 2 = A little bit 3 = Somewhat 4 = Quite a bit 5 = Very much |
| 15 | PA044 | In the past 7 days: | I felt content. | 1 = Not at all 2 = A little bit 3 = Somewhat 4 = Quite a bit 5 = Very much |

### General Life Satisfaction

| | | ( | General Life Satisfaction | |
|---|---|---|---|---|
| | Item ID | | For the next set of questions, please indicate how much you agree or disagree with each statement. | |
| 35 | PA045m | Indicate how much you agree or disagree: | In most ways, my life is close to perfect. | 1 = Strongly disagree 2 = Disagree 3 = Slightly disagree 4 = Neither agree nor disagree 5 = Slightly agree 6 = Agree 7 = Strongly agree |
| 36 | PA046 | Indicate how much you agree or disagree: | If I could live my life over, I would change almost nothing. | 1 = Strongly disagree 2 = Disagree 3 = Slightly disagree 4 = Neither agree nor disagree 5 = Slightly agree 6 = Agree 7 = Strongly agree |
| 37 | PA047 | Indicate how much you agree or disagree: | I am satisfied with my life. | 1 = Strongly disagree 2 = Disagree 3 = Slightly disagree 4 = Neither agree nor disagree 5 = Slightly agree 6 = Agree 7 = Strongly agree |
| 38 | PA048 | Indicate how much you agree or disagree: | So far I have gotten the important things I want in life. | 1 = Strongly disagree 2 = Disagree 3 = Slightly disagree 4 = Neither agree nor disagree 5 = Slightly agree 6 = Agree 7 = Strongly agree |
| 39 | PA049m | Indicate how much you agree or disagree: | My life situation is excellent. | 1 = Strongly disagree 2 = Disagree 3 = Slightly disagree 4 = Neither agree nor disagree 5 = Slightly agree 6 = Agree 7 = Strongly agree |

### **Meaning and Purpose**

| | | Strongly<br>disagree | Disagree | Neither<br>agree nor<br>disagree | Agree | Strongly<br>agree |
|---|---|---|---|---|---|---|
| PA203_<br>C | I have a good sense of what makes my life meaningful. | | | _ | | |
| PA205_<br>C | I generally feel that<br>what I do in my life is<br>valuable and<br>worthwhile. | | | | | |
| PA210_<br>C | I have very clear goals and aims for my life. | | | | | |

### Not at all A little bit Somewhat Quite a bit Very much

| | • | · <u> </u> | , , ,,,,,,, | <br><u> </u> | vory maor |
|---|---|---|---|---|---|
| PA221_<br>C | My life has meaning. | | | | |
| PA224_<br>C | My life has significance. | | | | |
| PA227_<br>C | I have a clear sense of direction in life. | | | | |
| PA232_<br>C | I experience deep fulfillment in my life. | | | _ | |
| PA237_<br>C | My life has purpose. | | | | |

### **General Self-Efficacy**

For the next set of questions, please read each sentence and rate your level of confidence in managing various situations, problems, and events.

| | | I am not<br>At all<br>Confident | I am a<br>a little<br>confident | I am<br>somewhat<br>confident | I am<br>quite<br>confident | I am very<br>confident |
|---|---|---|---|---|---|---|
| GSE11_C | I can manage to solve difficult problems if I try hard enough. | | | _ | | |
| GSE14_C | I am confident that I could deal efficiently with unexpected events. | | | | | |
| GSE19_C | If I am in trouble, I can think of a solution. | | | | | |
| GSE20_C | I can handle whatever comes my way. | | | | | |

# PROMIS-29 (+4 additional PROMIS physical functioning items and PROMIS Anger SF)

### Please respond to each question or statement by marking one box per row.

| | Physical Function | Without<br>any<br>difficulty | With a<br>little<br>difficulty | With<br>some<br>difficulty | With<br>much<br>difficulty | Unable<br>to do |
|---|---|---|---|---|---|---|
| 1 | Are you able to do chores such as vacuuming or yard work? | | | | | |
| 2 | Are you able to go up and down stairs at a normal pace? | | | | | |
| 3 | Are you able to go for a walk of at least 15 minutes? | | | | | |
| 4 | Are you able to run errands and shop? | | | | | |
| | | Not at all | Very little | Somewhat | Quite a lot | Cannot do |
| 5 | Does your health now limit you in doing two hours of physical labor? | | | | | |
| 6 | Does your health now limit you in doing moderate work around the house like vacuuming, sweeping floors or carrying in groceries? | | | | | |
| 7 | Does your health now limit you in lifting or carrying groceries? | | | | | |
| 8 | Does your health now limit you in doing heavy work around the house like scrubbing floors, or lifting or moving heavy furniture? | | | | | |
| | Anxiety In the past 7 days | Never | Rarely | Sometimes | Often | Always |
| 9 | I felt fearful | | | | | |
| 10 | I found it hard to focus on anything other than my anxiety | | | | | |
| 11 | My worries overwhelmed me | | | | | |
| 12 | I felt uneasy | | | | | |

| | Depression In the past 7 days | Never | Rarely | Sometimes | Often | Always |
|---|---|---|---|---|---|---|
| 13 | I felt worthless | | | | | |
| 14 | I felt helpless | | | | | |
| 15 | I felt depressed | | | | | |
| 16 | I felt hopeless | | | | | |
| | Anger During the past 7 days | Never | Rarely | Sometimes | Often | Always |
| 17 | I was irritated more than people knew | | | | | |
| 18 | I felt angry | | | | | |
| 19 | I felt like I was ready to explode | | | | | |
| 20 | I felt grouchy | | | | | |
| 21 | I felt annoyed | | | | | |
| | Fatigue During the past 7 days | Not at all | A little bit | Somewhat | Quite a bit | Very much |
| 22 | I feel fatigued | | | | | |
| 23 | I have trouble <u>starting</u> things because I am tired | | | | | |

| | Fatigue In the past 7 days | Not at all | A little bit | Somewhat | Quite a bit | Very much |
|---|---|---|---|---|---|---|
| 24 | How run-down did you feel on average? | | | | | |
| 25 | How fatigued were you on average? | | | | | |
| | Sleep Disturbance In the past 7 days | Very poor | Poor | Fair | Good | Very good |
| 26 | My sleep quality was | | | | | |
| | In the past 7 days | Not at all | A little bit | Somewhat | Quite a bit | Very much |
| 27 | My sleep was refreshing | | | | | |
| 28 | I had a problem with my sleep | | | | | |
| 29 | I had difficulty falling asleep | | | | | |
| | Ability to Participate in Social Roles and Activities | Never | Rarely | Sometimes | Usually | Always |
| 30 | I have trouble doing all of my regular leisure activities with others | | | | | |
| 31 | I have trouble doing all of the family activities that I want to do | | | | | |
| 32 | I have trouble doing all of my usual work (include work at home) | | | | | |
| 33 | I have trouble doing all of the activities with friends that I want to do | | | | | |
| | Pain Interference In the past 7 days | Not at all | A little bit | Somewhat | Quite a bit | Very much |
| 34 | How much did pain interfere with your day to day activities? | | | | | |
| 35 | How much did pain interfere with work around the home? | | | | | |
| 36 | How much did pain interfere with your ability to participate in social activities?. | | | | | |

### **PROMIS Global Items**

Please respond to each item by marking one box per row.

| | | Excellent | Very<br>good | Good | Fair | Poor |
|---|---|---|---|---|---|---|
| 5lob <b>a</b> 101 | In general, would you say your health is: | 5 | 4 | 3 | 2 | 1 |
| Slobal02 | In general, would you say your quality of life is: | 5 | 4 | 3 | 2 | 1 |
| Sloba 103 | In general, how would you rate your physical health? | 5 | □<br>4 | 3 | 2 | 1 |
| Sloba 104 | In general, how would you rate your mental health, including your mood and your ability to think? | 5 | | 3 | 2 | |
| Sloba 105 | In general, how would you rate your satisfaction with your social activities and relationships? | 5 | | 3 | 2 | |
| Sloba 109 | In general, please rate how well you carry out your usual social activities and roles. (This includes activities at home, at work and in your community, and responsibilities as a parent, child, spouse, employee, friend, etc.) | 5 | 4 | 3 | 2 | 1 |

| Global10 | How often have you been bothered by emotional problems such as feeling anxious, depressed or irritable? | 1 | 2 | 3 | 4 | 5 |
|---|---|---|---|---|---|---|
| Global08 | How would you rate your fatigue on average? | 1 | 2 | 3 | 4 | 5 |
| Global07 | How would you rate your pain on average? 0 1 2 No pain | 3 4 | 5 | 6 7 | 8 9 | 10<br>Worst<br>imaginable<br>pain |

#### Diet

- 1. About how many cups of fruit (including 100% pure fruit juice) do you eat or drink each day?
  - a. None
  - b. ½ cup or less
  - c. ½ cup to 1 cup
  - d. 1 to 2 cups
  - e. 2 to 3 cups
  - f. 3 to 4 cups
  - g. 4 or more cups

- 1 cup of fruit could be:
- 1 small apple
- 1 large banana
- 1 large orange
- 8 large strawberries
- 1 medium pear
- 2 large plums
- 32 seedless grapes
- 1 cup (8 oz.) fruit juice
- ½ cup dried fruit
- 1 inch-thick wedge of watermelon
- 2. About how many cups of vegetables (including 100% pure vegetable juice) do you eat or drink each day?
  - a. None
  - b. ½ cup or less
  - c. ½ cup to 1 cup
  - d. 1 to 2 cups
  - e. 2 to 3 cups
  - f. 3 to 4 cups
  - g. 4 or more cups

- 1 cup of vegetables could be:
- 3 broccoli spears
- 1 cup cooked leafy greens
- 2 cups lettuce or raw greens
- 12 baby carrots
- 1 medium potato
- 1 large sweet potato
- 1 large ear of corn
- 1 large raw tomato
- 2 large celery sticks
- 1 cup of cooked beans
- 3. About how often do you drink regular pop/soda or other sugar sweetened beverages (not diet or calorie-free) in a typical week?
  - a. Every day
  - b. 5 6 days a week
  - c. 3 4 days a week
  - d. 1 2 days a week
  - e. Less often than 1 day a week
  - f. I don't drink any regular soda/pop or other sugar sweetened beverages
- 4. How many times per week do you eat fast food meals or snacks?
  - a. Every day
  - b. 5 6 days a week

- c. 3 4 days a week
- d. 1 2 days a week
- e. Less often than 1 day a week
- f. I don't drink eat any fast food meals or snacks

| <u>Alcohol</u> | |
|---|---|
| 5. Do you drink alcohol? | ☐ Yes ☐ No |
| a. If yes, how many days per week do you drink alcohol? | |
| b. How many drinks containing alcohol do you have on a typical day<br>when you are drinking? | |
| Smoking | |
| 6. Do you currently smoke? | □ Yes □ No |
| a. If yes, how many packs a day do you smoke? | <del></del> |
| 7. Did you smoke previously? | □ Yes □ No |
| a. If you are a former smoker, how many years has it been since you quit? | |

### **Current Physical Activity**

For this questionnaire, we want you to recall your <u>current</u> leisure time physical activity (do not include work or household activities) during a **typical week**. When considering the number of times per week, please only include those times that you were physically active for **more than 15 minutes**.

| Exa | ample: You typically swim vigorously for 20 minutes 2 times ek: | per week and run for 4 | 0 minutes 3 times per |
|---|---|---|---|
| | | Times per Week | Average Duration Each<br>Time You Exercised (in<br>minutes) |
| 1) | Strenuous Exercise (Heart Beats Rapidly) (e.g., running, jogging, hockey, football, soccer, squash, basketball, cross country skiing, judo, roller skating, vigorous swimming, vigorous long distance bicycling) | <u> </u> | |
| | | Times per Week | Average Duration Each<br>Time You Exercised (in<br>minutes) |
| 1) | <b>Strenuous Exercise</b> (Heart Beats Rapidly) (e.g., running, jogging, hockey, football, soccer, squash, basketball, cross country skiing, judo, roller skating, vigorous swimming, vigorous long distance bicycling) | | |
| 2) | <b>Moderate Exercise</b> (Not Exhausting) (e.g., fast walking, baseball, tennis, easy bicycling, volleyball, badminton, easy swimming, alpine skiing, popular and folk dancing) | | |
| 3) | Mild Exercise (Minimal Effort) (e.g., yoga, archery, fishing from river bank, bowling, horseshoes, golf, snowmobiling, easy walking, | | |

| Date: | | | | | | | | 1.D. | # | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | Interv | ention | Evalu | ation ( | Phone | Interv | | | |
| Thank you for<br>telephone con<br>conversation<br>of RA] as a re | versat<br>will be | ion is be brief, | eing reunder 3 | corded t<br>0 minut | for qual<br>es. The | ity assu<br>en in on | rance p | urposes<br>1 you'll | . I expe | |
| ***** | **** | ***** | ***** | ***** | ***** | ***** | ***** | ***** | ***** | ******* |
| First, I'd like | to ask | you a f | ew que | stions a | bout the | ese sess | ions and | d the stu | ıdy so f | ar. |
| Let's go back | throug | gh the s | kills w | e've cov | ered: | | | | | |
| 1. Please | c. Gr<br>d. Fo<br>e. Inf<br>f. Pos<br>g. Pe<br>h. Go<br>i. Act | atitude<br>rmal M<br>Formal I<br>sitive R<br>rsonal s<br>pals<br>ts of Ki | Journal<br>lindfulr<br>Mindfu<br>Leappra<br>strength | ness (bro<br>lness (n<br>isal<br>ns | eath awa | areness<br>ess in o | )<br>daily life | | avorite | (9): |
| | | | | tive Eve | | | (_) | | | (-)- |
| | | | _ | italizing | | | | | | |
| | | | | itude Jo | | | | | | |
| | | | Min | dfulness | s Forma | l (Brea | th Awar | eness) | | |
| | | | Min | dfulness | s Inform | ıal (Miı | ndfulnes | ss in Da | ily Acti | vities) |
| | | | Posi | tive Rea | appraisa | .1 | | | | |
| | | | Pers | onal str | engths | | | | | |
| | | | Atta | inable ( | Goals | | | | | |
| | | | Acts | of Kin | dness | | | | | |
| what | extent | would | | comme | _ | | ly not" i<br>s to a fri | | eing "d | efinitely yes", to |
| 0<br>Definitely no | 1<br>t | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>Definitely |

| | | hat extent would ged with cancer? | • | | on to someon | e newly |
|---|---|---|---|---|---|---|
| De | 0 1<br>finitely not | 2 3 | 4 5 | 6 7 8 | 8 9 | 10<br>Definitely |
| * | ****** | ******* | ****** | ****** | ***** | ****** |
| Ho | | you to practice the your response) | e following ski | lls over the next ( | 6 months? | |
| 4. | Positive | Event: | | | | |
| | 0<br>Not at all | 1<br>Once a month | 2<br>Once a week | 3<br>2-3 times/week | 4<br>Daily | Other |
| 5. | Capitaliz | zing: | | | | |
| | 0<br>Not at all | 1<br>Once a month | 2<br>Once a week | 3<br>2-3 times/week | 4<br>Daily | Other |
| 6. | Gratitud | le Journal: | | | | |
| | 0<br>Not at all | 1<br>Once a month | 2<br>Once a week | 3<br>2-3 times/week | 4<br>Daily | Other |
| 7. | Mindful | Breath Awarene | ss: | | | |
| | 0<br>Not at all | 1<br>Once a month | 2<br>Once a week | 3<br>2-3 times/week | 4<br>Daily | Other |
| 8. | Mindful | ness in Daily Acti | vities: | | | |
| | 0<br>Not at all | 1<br>Once a month | 2<br>Once a week | 3<br>2-3 times/week | 4<br>Daily | Other |

| 9. | Positive | Reappraisal: | | | | |
|---|---|---|---|---|---|---|
| | 0 | 1 | 2 | 3 | 4 | Other |
| | Not at all | Once a month | Once a week | 2-3 times/week | Daily | |
| 10. | Personal | Strengths: | | | | |
| | 0 | 1 | 2 | 3 | 4 | Other |
| | Not at all | Once a month | Once a week | 2-3 times/week | Daily | |
| 11. | Attainab | le Goals: | | | | |
| | 0 | 1 | 2 | 3 | 4 | Other |
| | Not at all | Once a month | Once a week | 2-3 times/week | Daily | |
| 12. | Acts of I | Kindness | | | | |
| | 0 | 1 | 2 | 3 | 4 | Other |
| | Not at all | Once a month | Once a week | 2-3 times/week | Daily | |
| *** | ****** | | | ****** | ****** | ****** |
| | | Pla | anning for cont | inued practice | | |
| Foi | premise of Again the | of these coping ski<br>ese skills are like r | lls is that they on the conscience of the constant of the cons | d practice of the sk<br>only work if you con<br>don't exercise them<br>to you, you need to | ntinue to pra<br>, they aren't | ctice them.<br>likely to work |
| It | frequentl<br>practice l | y) but are less like ess). First let's ta | ly to continue (lk about the one | n above participant<br>XX skill from abov<br>that you plan to co<br>t into your day and | e participant<br>ntinue. Wha | is going to at about it is |

How about your least favorite skill? Can you tell me what about that one makes you less likely to try and incorporate it into your life?

| One of | the interesting things about any new skill is that after a while you might get bored with it |
|---|---|
| | or it may stop having the same impact that it had initially. If (skill participant rates as |
| | most likely to continue) starts getting old for you, you should go back to the skills and |
| | choose another one and increase your practice of that one. Let's talk about (XX skill that |
| | participant rated the second most likely to practice) and ways you might be able to |
| | incorporate that into your daily life. |

\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*\*

#### Questions about website usage:

Can you talk about your experience using the intervention website?

Probe: What features did you like?

What could have been clearer?

What did you think of the at home practice exercises?

*If the participant did not progress through all the lessons* Why did you stop at lesson X?

In about four weeks (cite specific dates), I will email you the final online questionnaire for the study. This will mark the end of your participation in the study.

Are there any questions I can answer for you now?

Thank you again for your time and participation in this study. We really appreciate it!

Hang up.